CLINICAL TRIAL: NCT01092429
Title: 2D and Tissue Doppler Imaging Echocardiography Analysis of Left Ventricular Regional Wall Motion and Prognosis
Acronym: TDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 96-1504B
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- one,two,and three vessels disease; mortality

SUMMARY:
Development of myocardial ischemia, and/or myocarditis would induce different changes in myocardial contraction behavior pattern,which maybe very subtle, and may not be detected by the 2D and m-mode echocardiography examinations. According to tissue Doppler imaging(TDI), they can be depicted by different models of echo with higher frame rates. In addition, many studies using TDI have significantly contributed of efforts to evaluate systolic and diastolic function and prognosis.

This study assess the value of the indices of left ventricular function obtained by using TDI in patient with coronary artery disease(CAD). We hypothesized that TDI will add incremental value for regional wall motion abnormality of CAD and its prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Angina
2. Acue coronary syndrome
3. Left ventricular systolic dysfunction

Exclusion Criteria:

1. Significant valvular disease
2. Active cancer status
3. Acute Renal failure
4. Contrast allergy history
5. Pregnancy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Accoring to recommendation of ACC/AHA, patient had classI indication to perform coronary angiography
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Gung Memorial Hospital at Linkou, Taipei, Taiwan